CLINICAL TRIAL: NCT04273750
Title: RAI & HRS: Relationship Between Relative Adrenal Insufficiency and Failure of Treatment in Hepatorenal Syndrome: A Prospective Pilot Study
Brief Title: RAI & HRS: Relationship Between Relative Adrenal Insufficiency and Failure of Treatment in Hepatorenal Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17/P/152
Record Dates: First submitted 2019-08-29; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2019-08

CONDITIONS: Liver Cirrhosis; Acute Kidney Injury; Hepato-Renal Syndrome
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury; Hepatorenal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Plasma renin activity: 0,5 mL of plasma EDTA
  * Plasma norepinephrine: 1,3 mL of plasma EDTA
  * Aldosterone: 0,5 mL of serum
  * TNF-alpha: 0,5 mL of serum
  * Interleukin-6: 0,3 mL of serum
  * Interleukin-10: 0,3 mL of serum
  * Interleukin-12: 0,5 mL of serum
  * 10 ml of urine will be centrifuged at 3000 rpm for 10 minutes at 4°C and storage specimens at - 80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatorenal syndrome is a life-threatening medical condition and a serious complication of advanced liver scarring (cirrhosis). It consists of a deterioration of the function of the kidneys caused by a severe alteration in the circulation (blood flow to the kidneys) due to liver cirrhosis. Only around half of the patients respond to treatment which consists of intravenous medication. Moreover, the adrenal glands, which are located on the kidneys, also suffer an alteration in the blood flow leading to deterioration in their function as well. Thus, these patients produced less cortisol than needed; this situation is called "relative adrenal insufficiency". Cortisol is an important hormone necessary in extreme situations such as severe diseases. This is a study which will assess the relationship between the presence of adrenal dysfunction and failure to treatment in patients with hepatorenal syndrome.

DETAILED DESCRIPTION:
This is a prospective, observational, descriptive, clinical study.

This is a single centre study. All patients admitted to the South West Liver Unit with decompensated cirrhosis will be screened according to their serum creatinine (sCr) level taken as part of standard of care at admission or during their hospitalization.

All patients with AKI stage 2-3 or with stage 1 and serum Creatinine >133 µmol/L who give consent to participate or consent is given by legal representative. Patients should meet all the inclusion criteria and none exclusion criteria.

The consent can be received by a medical doctor or by a research nurse involved in the study. The details will be recorded on the study delegation log.

Patients will be followed up during admission. Decompensation episodes including development of hepatic encephalopathy, worsening ascites, jaundice, GI bleeding related to portal hypertension, and infections will be recorded during follow up. Follow up finishes when the patient is discharged.

AKI is defined as an increase of at least 26 µmol/L or a percentage increase of at least 50% from baseline sCr value, within 48 hours. Baseline value should have occurred within the previous 7 days. When baseline sCr is not known investigators diagnose AKI when sCr is higher than 106 µmol/L.

All patients with AKI will have the following tests taken at admission or when they develop AKI, as per standard of care: Full blood count; electrolytes; liver profile including bilirubin, GGT, ALP, AST, and ALT; coagulation screen including PT, INR and APTT; C-reactive protein; blood cultures; glucose; bone profile, including phosphate and calcium.

Stages of AKI are defined as:

* Stage 1: increase of sCr ≥26 μmol/L or an increase in sCr ≥1.5-fold to 2-fold from baseline. When baseline value is not known, sCr>106 μmol/L.
* Stage 2: increase of sCr >2-fold to 3-fold from baseline. When baseline value is not known, sCr>176 μmol/L.
* Stage 3: increase of sCr >3-fold from baseline or sCr ≥353 μmol/L or initiation of renal replacement therapy. When baseline value is not known, sCr>353 μmol/L.

Investigators will include a participant when they are diagnosed with AKI stage 2 or 3 or with AKI stage 1 with persistent sCr >133 µmol/despite initial measures, then baseline blood samples and urine sample will be taken and short synacthen test (SST) will be performed as per standard of care. SST consists of taking a sample for baseline total cortisol followed by intravenous administration of 250 µg of corticotropin followed by a new sample taken 60 minutes later to test peak total cortisol.

Extra blood samples will be taken when the patient is included and they include: plasma renin activity, aldosterone, vasopressin, norepinephrine, tumour necrosis factor-alpha, Interleukin-6, Interleukin-12, Interleukin-10, blood sample for detection of bacterial DNA, urinary sample to detect neutrophil gelatinase-associated lipocalin (NGAL).

Samples should be taken within 48 hours of diagnosis of AKI and always before treatment with terlipressin is started.

Patients will be managed according to our local guidelines and national and international standards. Human albumin (HAS) will be administered at 1 gram per Kilogram of weight in those participants with AKI stage 2-3 or those with AKI stage 1 who do not improve or progress. If there is no response after 48 hours of administration of HAS and HRS criteria are met, then vasoconstrictor treatment with terlipressin will be started.

Response to treatment is defined as a reduction of at least 25% from pre-treatment value. Full response is met when sCr returns to a value lower than 26 μmol/L above the baseline value. Partial response is met when final sCr returns to a value higher than 26 μmol/L above the baseline value.

During hospitalization vital signs and standard liver and renal tests will be recorded.

All interventions and follow-up will be carried out during the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects capable of giving informed consent, or in case of lack of capacity, their legal representative consent on their behalf.
* Older than 18 years old and younger than 80 years old.
* Diagnosis of cirrhosis according to liver biopsy, or non-invasive markers (Fibroscan) or a combination of clinical and imaging criteria.
* Diagnosis of AKI stage 2-3 or stage 1 with serum Creatinine > 133 µmol/L, according to the last international consensus (International Club of Ascites, 2015)

Exclusion Criteria:

* Advanced hepatocellular carcinoma, Barcelona-Clinic liver cancer (BCLC) stage C or D
* Infection by human immunodeficiency virus (HIV)
* Previous transplant or any other type of immunodeficiency
* Pregnancy
* Long-term treatment with steroids or other immunosuppressive agents or interferon
* Severe chronic heart failure, New York Heart Association (NYHA), class III or IV
* Advanced COPD, global initiative for chronic obstructive lung disease (GOLD) III or IV
* Renal failure on haemodialysis
* Any medical condition that gives a survival shorter than 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatorenal syndrome is a life-threatening medical condition and a serious complication of advanced liver scarring (cirrhosis). It consists of a deterioration in the function of the kidneys caused by a severe alteration in the blood flow to the kidneys due to liver cirrhosis. Around half of patients respond to treatment. The adrenal glands (located on the kidneys), suffer a variation in blood flow leading to deterioration in their function. Thus these patients produce less cortisol than needed; this situation is called "relative adrenal insufficiency". Cortisol is an important hormone necessary in extreme situations such as severe diseases. This study is to assess the relationship between the presence of adrenal dysfunction and failure to treatment in patients with hepatorenal syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Response to treatment | Between days 5 to 14 after treatment has started
  Reduction in sCr with terlipressin in patients with hepatorenal syndrome between patients with and without relative adrenal insufficiency. ** Definition of response to treatment: Response to treatment is defined as a reduction of at least 25% from pre-treatment value. Full response is met when final sCr returns to a value lower than 26 µmol/L above the baseline value. Partial response is met when final sCr returns to a value higher than 26 µmol/L above the baseline value. Always with a reduction of sCr of at least 25% from pre-treatment value.

SECONDARY OUTCOMES:
Hospital Mortality Rates | Through study completion an average of 20 months
  Hospital survival in patients with RAI and HRS. It's expected that patients with RAI and HRS have a higher mortality rate.
Bacterial Translocation | At baseline
  Association between bacterial translocation and RAI and response to treatment of hepatorenal syndrome.
Degree of Inflammation | At baseline
  Association between degree of inflammation (as measured by inflammatory markers) and response to treatment of hepatorenal syndrome.
Circulatory Dysfunction | At baseline
  Association between circulatory dysfunction and response to treatment in hepatorenal syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Acevedo, MD, Principal Investigator — jacevedo@nhs.net
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom